CLINICAL TRIAL: NCT02577809
Title: An Investigation of the Influence of Different Intrathecal Opioids on the Post-operative Pain Experiences of Woman at Rahima Moosa Mother and Child Hospital
Brief Title: Intrathecal Opioid Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Sean Chetty, Senior Clinical Lecturer, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M141181
Record Dates: First submitted 2015-10-10; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Fentanyl; Indomethacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Morphine100 (Active Comparator): 1.8ml 0.5% hyperbaric bupivacaine with 0.1mg preservative-free morphine (mixed in 0.4ml normal saline to a volume of 2.3ml) administered into the intrathecal space
  Interventions: Drug: Morphine100; Drug: Hyperbaric Bupivicaine; Drug: Indomethacin
- Morphine50 (Active Comparator): 1.8ml 0.5% hyperbaric bupivacaine with 0.05mg preservative-free morphine (mixed in 0.4ml normal saline to a volume of 2.3ml) administered into the intrathecal space
  Interventions: Drug: Morphine50; Drug: Hyperbaric Bupivicaine; Drug: Indomethacin
- Fentanyl25 (Active Comparator): 1.8ml 0.5% hyperbaric bupivacaine with 25μg fentanyl (2.3ml volume) administered into the intrathecal space
  Interventions: Drug: Fentanyl; Drug: Hyperbaric Bupivicaine; Drug: Indomethacin

INTERVENTIONS:
Drug: Morphine100 — 100mcg added to the spinal anaesthetic
  Other Names: Morphine 100 mcg
  Arms: Morphine100
Drug: Morphine50 — 50mcg added to the spinal anaesthetic
  Other Names: Morphine 50mcg
  Arms: Morphine50
Drug: Fentanyl — 25mcg Fentanyl added to the spinal anaesthetic
  Other Names: Fentanyl 25mcg
  Arms: Fentanyl25
Drug: Hyperbaric Bupivicaine — 1.8ml 0.5% spinal bupivicaine with dextrose
  Other Names: Spinal Bupivicaine
Drug: Indomethacin — 100mg Indomethacin suppository
  Other Names: Indomethacin Suppository

SUMMARY:
This is an interventional drug trail to evaluate the effect of different intrathecal opioids on post-operative pain experiences in women who have undergone caesarean section surgery.

DETAILED DESCRIPTION:
1. To evaluate the effect of three different intrathecal opioid mixtures on post-operative pain experiences in women who have undergone caesarean section surgery, relating specifically to:

   1. Post-operative analgesic requirements at two time points (12 hours and 24 hours) after surgery
   2. Pain scores at two time points (12 hours and 24 hours) after surgery
   3. Sedation scores at two time points (12 hours and 24 hours) after surgery
   4. Post-operative nausea scores at two time points (12 hours and 24 hours) after surgery
   5. Post-operative pruritis scores at two time points (12 hours and 24 hours) after surgery
2. To determine the impact that the patients' post-operative pain has on their activities in the first 24 hours after surgery

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18years having caesarean section surgery under single shot spinal neuraxial anaesthesia at Rahima Moosa Mother and Child Hospital

Exclusion Criteria:

* Pre-operative:

  b) Patient refusal or inability to give informed consent c) Severe pre-eclampsia d) Eclampsia e) Patient unable to understand how to use the Patient Controlled Analgesia (PCA) pump, after appropriate counselling and training
* Intra-operative:

  a) Obstetric Complications: i) Post-partum Haemorrhage ii) Ruptured Uterus iii) Still Birth b) Conversion to general anaesthesia intra-operatively c) Administration of supplementary intravenous opioid analgesics
* Post-operative:

  1. Patients who have babies that require additional care, for a prolonged period, after birth eg. Neonatal ICU admission for ≥ 12hours or congenital abnormalities
  2. Patients who require ICU or High care admission postoperatively for any intra-operative complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Opioid Analgesic Requirements measured by total morphine usage on Patient Controlled Analgesic pump | For 24 hours after surgery
  The total administered morphine dose administered to the patient through the PCA pump will be documented. This is documented at 24 hours after surgery.
Patient Pain Score measured by the Numeric Pain Rating scale | 24 hours after surgery
  The instrument consists of 11 numbered points ( 0 to 10) each of which represent a different pain level for the patient. The scale ranges from 0=NO PAIN up to 10= worst pain possible. This is assessed at 24 hours after surgery.
Patient sedation scores measured by a 4 point sedation scale | 24 hours
  The instrument consists of 4 numbered points ( 0 to 3) each of which represent a different level of sedation for the patient. The scale ranges as follows: 0 =awake, 1 = mild drowsiness, 2 = moderate drowsiness, easily awaken, 3 =difficult to arouse.This is assessed at 24 hours after surgery.
Patient post-operative nausea and vomiting score using a 4 point scale | 24 hours
  The instrument consists of 4 numbered points ( 0 to 3) each of which represent a different level of nausea for the patient. The scale ranges as follows: 0 = No Nausea, 1 = presence of nausea without vomiting, 2 = mild to moderate vomiting (not requiring treatment), 3 = severe vomiting (treatment required). This is assessed at 24 hours after surgery.
Patient post-operative pruritis Score using a 2 point scale | 24 hours
  The instrument consists of 3 numbered points ( 0 to 2) each of which represent a different level of pruritus for the patient. The scale ranges as follows: 0 = no pruritus, 1 = mild to moderate pruritus (not requiring treatment), 2 = severe pruritus (treatment required). This is assessed at 24 hours after surgery.
Patient respiratory rate measured by counting the respiratory rate over a one minute period | 24 hours
  The patients respiratory rate will be counted by the investigator at the time of evaluation at 24hours after surgery. The resulted will be documented as a rate per minute.

SECONDARY OUTCOMES:
The Impact of the patients pain on their activity measured using an 11 point scale | 24 hours
  The instrument consists of 11 numbered points ( 0 to 10) each of which represent a different levels of interference with the patients activity since surgery. The scale ranges from 0= DID NOT INTERFERE up to 10= COMPLETELY INTERFERED. This is assessed at 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Chetty, FCA(SA), Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Rahima Moosa Mother and Child Hospital, Johannesburg, Gauteng, South Africa